CLINICAL TRIAL: NCT06153134
Title: Effectiveness of Curcuma Xanthorriza Roxb. 10% Cream in Reducing Melasma Area and Severity Index (MASI) Scores and Improvement of Skin Brightness in Epidermal Type Melasma
Brief Title: Curcuma Xanthorriza Roxb. 10% Cream for Melasma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DV-202311.01
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Melasma
Keywords: Melasma; MASI; Specthrophotometry; Curcuma xanthorriza; Curcuma; Depigmenting agent
MeSH Terms: conditions — Melanosis | interventions — kojic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcuma xanthorriza Roxb. (Active Comparator): Fifteen patients will apply 10% Curcuma xanthorriza Roxb. cream topically at the half of the face, once daily in night, for 2 months.
  Along with study drug or positive control, patients will receive standard uniform sunscreen and face wash.
  Interventions: Drug: 10% Curcuma xanthorriza Roxb.
- Kojic acid (Active Comparator): Fifteen patients will apply 2% kojic acid cream topically at the half of the face, once daily in night, for 2 months.
  Along with study drug or positive control, patients will receive standard uniform sunscreen and face wash.
  Interventions: Drug: 2% Kojic Acid

INTERVENTIONS:
Drug: 10% Curcuma xanthorriza Roxb. — Patients in experimental arms will receive 10% Curcuma xanthorriza Roxb. cream for 2 months
  Arms: Curcuma xanthorriza Roxb.
Drug: 2% Kojic Acid — Patients in experimental arms will receive 2% Kojic Acid cream for 2 months
  Arms: Kojic acid

SUMMARY:
Melasma is an acquired hyperpigmentation disorder with a multifactorial etiology and complex pathogenesis that can significantly diminish the quality of life for affected patients. As of now, melasma therapy remains challenging due to its high recurrence rate and the common occurrence of treatment-related side effects. The use of depigmentation agents is a crucial component in managing melasma. Hydroquinone stands as the first-line depigmentation agent for melasma; however, its use often leads to adverse effects. Therefore, alternative depigmentation agents are needed. Curcuma xanthorriza Roxb., a native plant of Indonesia, operates by inhibiting the tyrosinase enzyme, reducing MITF transcription, and inhibiting α-MSH. Despite these potential benefits, Curcuma xanthorriza Roxb. has not been utilized as a depigmentation agent. Research on the effectiveness of Curcuma xanthorriza Roxb. as a depigmentation agent in melasma treatment has not been conducted. Therefore, it is essential to conduct research to determine the effectiveness of a 10% Curcuma xanthorrhiza Roxb. cream in reducing MASI scores and enhancing skin brightness in epidermal-type melasma.

DETAILED DESCRIPTION:
Curcuma xanthorrhiza Roxb., known locally as temulawak in Indonesia or koneng gede in Sundanese, is a member of the Zingiberaceae family and is native to Indonesia. Previous research related to Curcuma xanthorriza Roxb. and its impact on melanin synthesis was conducted using mushroom tyrosinase by Batubara et al. The study found that methanol extract of Curcuma xanthorriza Roxb. could decrease tyrosinase enzyme activity with an inhibition concentration 50% (IC50) of 0.27 mg/mL.

Research conducted by Lee et al. on curcumin from another Curcuma species, C. longa or turmeric, demonstrated that curcumin reduced melanin quantity, tyrosinase enzyme activity, and micropthalmia-associated transcription factor (MITF) protein. In an in-silico study, Mustarichie et al. reported that the three active compounds in Curcuma xanthorriza Roxb. could inhibit both tyrosinase enzyme and α-melanin stimulating hormone (α-MSH). Xanthorrizol exhibited the most effective interaction with the tyrosinase enzyme, while demethoxycurcumin showed the most effective interaction with α-MSH.

Up to this point, there has been no research on the effectiveness of 10% Curcuma xanthorriza Roxb. cream in treating melasma. Therefore, the researchers are motivated to investigate the efficacy of 10% Curcuma xanthorriza Roxb. cream as a depigmentation agent, based on the assessment of MASI scores and skin brightness levels in patients with epidermal-type melasma using split-face therapy.

ELIGIBILITY:
Inclusion Criteria:

* Females and males diagnosed with epidermal-type melasma clinically and through Wood's lamp examination.
* Study subjects exhibit melasma lesions on both sides of the face.

Exclusion Criteria:

* History of hypersensitivity to Curcuma xanthorriza Roxb. or kojic acid based on anamnesis.
* Pregnant and breastfeeding women.
* Patients using hormonal contraceptive drugs in the last 3 months.
* Patients using topical medications (depigmentation agents, tretinoin, or corticosteroids) in the skin area to be tested in the last 2 weeks.
* Patients using systemic corticosteroids in the last 1 month.
* Patients undergoing laser therapy, microdermabrasion, chemical peels, and other aesthetic procedures in the skin area to be tested in the last 1 month.
* Patients experiencing inflammation on the facial skin.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-12-22 (Estimated); Primary Completion 2024-02-22 (Estimated); Study Completion 2024-05-22 (Estimated)

PRIMARY OUTCOMES:
Modified Melasma Area and Severity Index (MASI) score | 56 days
  Measurement scale for subjectively assessing the severity of melasma. There are three variables used to gauge the severity of melasma, namely darkness (D), homogeneity (H), and involved area (A).
Skin Brightness | 56 days
  The brightness level of the skin is measured using a spectrophotometer. Skin brightness is assessed based on the L* value, which ranges from total darkness (L* = 0) to total whiteness (L* = 100).

SECONDARY OUTCOMES:
Side Effects | 56 days
  Undesirable reactions that may occur on the skin following therapy with 10% Curcuma xanthorriza Roxb. cream or 2% kojic acid cream include sensations such as itching, a burning sensation, erythema, erythematous papules, edema, blistering, urticaria, or post-inflammatory hyperpigmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Reti Hindritiani, M.D., Study Chair — Faculty of Medicine Universitas Padjadjaran Bandung; Diah Puspitosari, M.D., Study Director — Faculty of Medicine Universitas Padjadjaran Bandung; Fathia Rianty, M.D., Study Director — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia